CLINICAL TRIAL: NCT00405782
Title: Pilot Study of a Moderate-Intensity Exercise Intervention in Women With Metastatic Breast Cancer
Brief Title: Exercise Intervention in Women With Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer A. Ligibel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06-212
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: metastatic breast cancer; exercise intervention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Exercise Group (Active Comparator): Exercise Intervention begins immediately
  Interventions: Behavioral: Moderate-Intensity Exercise
- Delayed Exercise Group (Active Comparator): Exercise intervention delayed by 16 weeks
  Interventions: Behavioral: Moderate-Intensity Exercise

INTERVENTIONS:
Behavioral: Moderate-Intensity Exercise — Exercise program designed by exercise physiologist

SUMMARY:
This study is being done to evaluate the impact of moderate-intensity exercise (such as walking) on quality of life, energy level, endurance and mood in women with metastatic breast cancer. Studies have shown that women with early stage breast cancer who exercise during treatment have more energy, less sleep disturbance, less anxiety and depression, and better strength and endurance than women who do not exercise. These studies have also shown that women who exercised during treatment for early stage breast cancer did not develop injuries or increased fatigue from exercising during chemotherapy and radiation treatments. The investigators are conducting this trial to see if women with metastatic breast cancer experience similar benefits from exercise as women with earlier breast cancer. The investigators also wish to determine whether women with advanced disease are able to exercise safely during their treatment under the supervision of an exercise physiologist.

DETAILED DESCRIPTION:
* Participants will be randomized to one of two groups. Study participants assigned to Group A will immediately participate in a 16-week exercise program, and participants assigned to Group B will wait 16 weeks before taking part in an exercise program.
* Before beginning the exercise program (Group A) or waiting period (Group B), participants will undergo a series of tests to measure exercise capacity, fatigue level and quality of life. They will be asked to complete a series of questionnaires and meet with an exercise physiologist and undergo a treadmill test designed to measure physical fitness in patients with a chronic illness. The participant will complete the questionnaires again 8 weeks after enrolling in the protocol and will complete one final set and undergo a second treadmill test after the 16-week study period has ended.
* Participants in Group A will be given a 16-week gym membership, as well as a heart rate monitor and a pedometer. They will meet with an exercise physiologist, who will design an exercise program for each participant. Participants will meet with the exercise physiologist weekly for 4 weeks, then once per month for the duration of the study. The target exercise goal will be 150 minutes of moderate-intensity exercise each week.
* Participants will be given an exercise journal to record the minutes of cardiovascular exercise and steps taken each day. These journals will be reviewed by the exercise physiologist each week.
* Participants in Group B will be allowed to exercise as much as they wish during the first 16-weeks of their time on the study, but they will not be given a formal exercise plan or a gym membership until the completion of the 16-week waiting period. During this time, they will also complete questionnaires at the time of study entry, 8 weeks after enrolling, and at the end of 16 weeks. After the 16-week delay period has passed, participants in Group B will be given a pedometer, heart rate monitor and 16-week gym membership. They will also meet with an exercise physiologist weekly for one month, and the exercise physiologist will design an individualized exercise plan for these participants.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally advanced breast cancer not amenable to curative surgery
* Life expectance of greater than 12 months
* English speaking
* Pre- and postmenopausal
* Performance status 0-1

Exclusion Criteria:

* Baseline exercise of more than 150 minutes/week
* Active brain metastases
* Uncontrolled cardiac disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-08; Primary Completion 2014-08 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To determine the impact of a 16 week exercise intervention on physical functioning and cardiorespiratory fitness in a group of patients with metastatic breast cancer. | 16 weeks

SECONDARY OUTCOMES:
To determine the impact of a 16-week exercise intervention on quality of life, fatigue and mood in a group of patients with metastatic breast cancer | 16 weeks
To test the feasibility of an exploratory measure of health care utilization in a population of patients with metastatic breast cancer and potential impact on a 16-week exercise intervention on health care utilization. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No